CLINICAL TRIAL: NCT02621723
Title: Capturing Readmission Internationally to Prevent Readmission by Safer@Home
Brief Title: Capturing Readmission Internationally to Prevent Readmission by Safer@Home Group
Acronym: CURIOS@
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Prabath W.B. Nanayakkara, PhD, MD, FRCP, Amsterdam UMC, location VUmc
Other Study IDs: VUMedicalcenter
Record Dates: First submitted 2015-11-25; First posted 2015-12-03 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Hospital Readmission
Keywords: Preventability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
CURIOS@ is a prospective multi-centre cross-sectional study to investigate readmissions in participating units. The data collected is derived from two clinical episodes: the episode containing the re-admission and the previous admission (index admission).

The main aims are:

Outcomes:

* Risk factors to predict preventable readmissions in non-surgical patients
* Percentage of subjectively non-preventable and preventable readmissions from patient, carer, their nurses and their physician's point of view
* Comparison for risk factors on readmissions throughout Europe
* Increasing awareness and knowledge for health-care workers on readmissions and its preventability

DETAILED DESCRIPTION:
Data will be derived directly from patients, from the clinical notes of the previous admission and records of discharge communication. Also information from treating physicians, nurses and immediate caregivers will be collected. The data set will contain no directly identifiable variables (data will be registered by using a research code for each patient).

Data collection will include: Hospital-related data, patient-related data, health-related data, time-related data, and physician related data. Also patient feedback is requested.

After obtaining written informed consent, the researcher will ask the patient 7 questions about the (preventability of their) readmission. Also the patient will be asked if one of the direct carers can be approached with 2 questions. The carer will most often be a sibling, a good friend or someone from the neighborhood. We will approach the carer in person or by telephone, and only after explicit permission from the patient. Lastly, we will ask a doctor and nurse (responsible for the patient in the first 24 hours of his readmission) similar questions.

ELIGIBILITY:
Inclusion criteria:

* Adult patients aged 18 or above admitted to hospital as unscheduled medical admission for a minimum of a single night following a previous admission within 30 days
* Index admission can be for any procedure (elective/non-elective)
* Index admission at any hospital ward (except psychiatry, pediatrics or gynaecology) for a minimum of a single night during the previous 30 days
* Readmission should be to a medical ward (Medical ward: Cardiology, geriatrics, gastroenterology, hematology, internal medicine, nephrology, neurology, oncology, pulmonary medicine, rheumatology.)
* If a patient is readmitted more than once within the study period, only the first readmission will be included
* The port of entry is through an Emergency Department, Acute Medical Unit or any other clinical ward (i.e. department of internal medicine).
* Patients should all be capable of understanding the study and give written informed consent. They should all be mentally competent.

Exclusion criteria:

* Patients readmitted electively for procedures, surgery or chemotherapy
* Patients readmitted for a non-medical specialism (surgery, urology, ent etc..)
* Patients admitted or readmitted who are pregnant
* Patients admitted or readmitted aged under 18
* Patients index or readmission for pediatrics, psychiatry, gynaecology
* Patients who stayed less than one night during index and readmission
* Patients who have been admitted to another institution in their index admission (To facilitate timely case identification and ready access to treating physicians, we will only review same-hospital readmissions)
* A second readmission for the same patient within the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients readmitted for at least one night for a medical specialism after any type of admission at any ward in the previous 30 days, with an overnight stay. This could be from any ward, for any procedure (elective/non-elective)
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of readmissions deemed preventable by patients, their informal carers, nurses and physicians | 1 year
  Of all the readmissions in the study, we will look at the readmissions which are deemed potentially preventable (YES or NO) by all partners of care chain. In the end this will give us a percentage of readmissions judged as potentially preventable by all partners of care chain.

SECONDARY OUTCOMES:
Causes of preventable readmissions | 1 year
  We will ask all partners in the care chain about the causes of the readmissions. These will be categorised:
  Disease-related: Natural progress disease, out of control/influence physician or patient - for example: metastasis cancer.
  Patient-related: Related to control/influence patient, out of control/influence professionals - for example: a patient who refused extra home care after the index admission.
  Human/caregiver-related: Related to the control/influence professionals - for example: poor medication handover after index inclusion.
  Organisational: Readmission related to organisational problems - for example: no beds available, transfer from other hospital etc.
  Technical: Readmission related to technical defects of materials or equipment - for example: IV-drip home infusion antibiotics broken.
Risk factors for preventable readmissions | 1 year
  For every readmission, we will ask researchers to fill out a dataset with potential risk factors. These are:
  1. General data regarding readmission: i.e. length of stay, time between index admission and readmission.
  2. Patient-related factors: i.e. age, sex, marital status, living situation etc.
  3. Health-related: ie. comorbiditity, frailty score, polypharmacy etc.
  4. Time-related: i.e. Total admissions in previous year
  5. Physician related: i.e. was a discharge letter send?

CONTACTS AND LOCATIONS:
Locations (8):
- Hospital of South West Jutland, Esbjerg, Denmark
- Netherlands (5):
  - VU University Medical Centre, Amsterdam, North Holland
  - Academic Medical Centre (AMC), Amsterdam
  - Albert Schweitzer, Dordrecht
  - Westfriesgasthuis, Hoorn
  - VieCuri Hospital, Venlo
- United Kingdom (2):
  - Ysbyty Gwynedd Hospital, Bangor
  - University Hospital of South Manchester, Manchester

REFERENCES:
- [Background] Greysen SR, Stijacic Cenzer I, Auerbach AD, Covinsky KE. Functional impairment and hospital readmission in Medicare seniors. JAMA Intern Med. 2015 Apr;175(4):559-65. doi: 10.1001/jamainternmed.2014.7756. PMID 25642907
- [Background] Zanocchi M, Maero B, Martinelli E, Cerrato F, Corsinovi L, Gonella M, Ponte E, Luppino A, Margolicci A, Molaschi M. Early re-hospitalization of elderly people discharged from a geriatric ward. Aging Clin Exp Res. 2006 Feb;18(1):63-9. doi: 10.1007/BF03324642. PMID 16608138
- [Background] Donze J, Aujesky D, Williams D, Schnipper JL. Potentially avoidable 30-day hospital readmissions in medical patients: derivation and validation of a prediction model. JAMA Intern Med. 2013 Apr 22;173(8):632-8. doi: 10.1001/jamainternmed.2013.3023. PMID 23529115
- [Background] van Walraven C, Wong J, Forster AJ. LACE+ index: extension of a validated index to predict early death or urgent readmission after hospital discharge using administrative data. Open Med. 2012 Jul 19;6(3):e80-90. Print 2012. PMID 23696773
- [Background] Drame M, Lang PO, Novella JL, Narbey D, Mahmoudi R, Laniece I, Somme D, Gauvain JB, Heitz D, Voisin T, de Wazieres B, Gonthier R, Ankri J, Saint-Jean O, Jeandel C, Couturier P, Blanchard F, Jolly D. Six-month outcome of elderly people hospitalized via the emergency department: the SAFES cohort. Rev Epidemiol Sante Publique. 2012 Jun;60(3):189-96. doi: 10.1016/j.respe.2011.11.004. Epub 2012 May 16. PMID 22608011
- [Background] Cooksley T, Nanayakkara PW, Nickel CH, Subbe CP, Kellett J, Kidney R, Merten H, Van Galen L, Henriksen DP, Lassen AT, Brabrand M; safer@home consortium. Readmissions of medical patients: an external validation of two existing prediction scores. QJM. 2016 Apr;109(4):245-8. doi: 10.1093/qjmed/hcv130. Epub 2015 Jul 10. PMID 26163662
- [Background] Hansen LO, Williams MV, Singer SJ. Perceptions of hospital safety climate and incidence of readmission. Health Serv Res. 2011 Apr;46(2):596-616. doi: 10.1111/j.1475-6773.2010.01204.x. Epub 2010 Nov 24. PMID 21105868
- [Background] Billings J, Blunt I, Steventon A, Georghiou T, Lewis G, Bardsley M. Development of a predictive model to identify inpatients at risk of re-admission within 30 days of discharge (PARR-30). BMJ Open. 2012 Aug 10;2(4):e001667. doi: 10.1136/bmjopen-2012-001667. Print 2012. PMID 22885591
- [Background] Jackson AH, Fireman E, Feigenbaum P, Neuwirth E, Kipnis P, Bellows J. Manual and automated methods for identifying potentially preventable readmissions: a comparison in a large healthcare system. BMC Med Inform Decis Mak. 2014 Apr 5;14:28. doi: 10.1186/1472-6947-14-28. PMID 24708889
- [Background] Davies S, Saynina O, Schultz E, McDonald KM, Baker LC. Implications of metric choice for common applications of readmission metrics. Health Serv Res. 2013 Dec;48(6 Pt 1):1978-95. doi: 10.1111/1475-6773.12075. Epub 2013 Jun 6. PMID 23742056
- [Background] Blunt I, Bardsley M, Grove A, Clarke A. Classifying emergency 30-day readmissions in England using routine hospital data 2004-2010: what is the scope for reduction? Emerg Med J. 2015 Jan;32(1):44-50. doi: 10.1136/emermed-2013-202531. Epub 2014 Mar 25. PMID 24668396
- [Background] Bianco A, Mole A, Nobile CG, Di Giuseppe G, Pileggi C, Angelillo IF. Hospital readmission prevalence and analysis of those potentially avoidable in southern Italy. PLoS One. 2012;7(11):e48263. doi: 10.1371/journal.pone.0048263. Epub 2012 Nov 2. PMID 23133624
- [Background] Cooksley T, Merten H, Kellett J, Brabrand M, Kidney R, Nickel CH, Nanayakkara PW, Subbe CP. PRISMA Analysis of 30 Day Readmissions to a Tertiary Cancer Hospital. Acute Med. 2015;14(2):53-6. PMID 26305081